CLINICAL TRIAL: NCT03715322
Title: Efficacy and Safety of Inhaled Tobramycin on Bronchiectasis Colonized With Pseudomonas Aeruginosa: A Randomized, Double-blind, Parallel-group Multicenter Trial
Brief Title: Tobramycin in Bronchiectasis Colonized With Pseudmonas Aeruginosa
Acronym: TORNASOL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, Associated professor; principal investigator (respiratory medicine), Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIRH-2018-TOBRA
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Bronchiectasis Adult; Pseudomonas Infections
Keywords: bronchiectasis; Pseudomonas aeruginosa; tobramycin; nebulization; bacterial load; quality of life
MeSH Terms: conditions — Pseudomonas Infections; Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into the treatment group and control group. No cross-over of the study group will be made.
Who Masked: Participant, Investigator
Masking Description: Both the investigators and the participants will be masked to the study allocation. The randonmization codes will be generated by a blinded medical statistician with the use of computerized program. Randomization will be achieved based on the permuted block design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tobramycin inhalation (Active Comparator): 300mg tobramycin dissolved in 5ml saline will be nebulized with an ultrasonic nebulizer within 15-20 minutes.
  Interventions: Drug: Tobramycin Inhalant Product; Other: usual care
- natural saline inhalation (Placebo Comparator): 5ml saline will be nebulized with an ultrasonic nebulizer within 15-20 minutes.
  Interventions: Other: usual care; Drug: Natural saline inhalation
- usual care (Other): ambroxool (30mg thrice daily), or N-acetylcysteine (0.2g thrice daily) plus chest physiotherapy (5 min, once daily)
  Interventions: Drug: Tobramycin Inhalant Product; Drug: Natural saline inhalation

INTERVENTIONS:
Drug: Tobramycin Inhalant Product — Tobramycin will be nebulized (300mg twice daily) with an ultrasonic nebulizer. A total of two 28-day on-and-off cycles will be scheduled.
  Arms: tobramycin inhalation; usual care
Other: usual care — ambroxool (30mg thrice daily), or N-acetylcysteine (0.2g thrice daily) plus chest physiotherapy (5 min, once daily)
  Arms: natural saline inhalation; tobramycin inhalation
Drug: Natural saline inhalation — Natural saline will be nebulized (5ml twice daily) with an ultrasonic nebulizer. A total of two 28-day on-and-off cycles will be scheduled.
  Arms: natural saline inhalation; usual care

SUMMARY:
This is a phase 3 study. Patients will be enrolled from 14 medical centers in mainland China. Eligible patients will be randomly allocated to treatment group (tobramycin nebulization, 300mg bid) and control group (natural saline nebulization, 5ml bid). A total of two 28-day on-and-off cycles will be scheduled. Both tobramycin solution and natural saline and the nebulizer will be solely provided by the sponsor.

DETAILED DESCRIPTION:
This is a phase 3 study. All bronchiectasis patients will be enrolled from 14 medical centers located in different geographic regions of mainland China. After a three-week screening period, On the basis of usual care [ambroxool (30mg thrice daily) or N-acetylcysteine (0.2g thrice daily) and chest physiotherapy (5 min, once daily)], eligible patients will be randomly allocated to treatment group (tobramycin nebulization, 300mg bid, delivered via an ultrasonic nebulizer) and control group (natural saline nebulization, 5ml bid, delivered via an ultrasonic nebulizer). A total of two 28-day on-and-off cycles will be scheduled. At the end of each on-and-off cycle, sputum culture and other clinical assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years, had a history of chronic cough and sputum production, had physician-diagnosed bronchiectasis based on high-resolution chest computed tomography (effective within 12 months)
* Remaining clinically stable (no significant changes in respiratory symptoms and free from upper respiratory tract infection or bronchiectasis exacerbations for 4 weeks)
* Sputum culture positive to Pseudomonas aeruginosa at screening
* Forced expiratory volume in one second > 30% predicted and < 80% predicted
* Could tolerate to nebulization
* At least one bronchiectasis exacerbation within the past two years
* Can correctly nebulize the study medications and fill in the diary cards following instruction of the investigators

Exclusion Criteria:

* Had a knwon history of allergy to tobramycin
* Had concomitant asthma, allergic bronchopulmonary aspergillosis, active tuberculosis, or active infection with non-tuyberculous mycobacteria that warranted regular anti-mycobacterial treatment
* Had moderate or major haemoptysis within 6 months
* Had concomitant severe cardiovascular diseases or haematopoietic diseases (congestive heart failure, clinically significant coronary heart disease, myocardial infarction or stroke, clinically arrythmia, known anurysm of the aorta, uncontroll hypertension (systolic blood pressure > 160mmHg or diastolic pressure >100mmHg at two consecutive time points)
* Concomitant severe psychiatric disorders
* Uncontrolled diabetes mellitus or fasting blood glucose >10mmol/L
* Active peptic or duodenal ulcer
* Moderate-to-severe gastroesophageal reflux diseases
* Malignancy
* Severe myasthenia gravis or Parkinson's disease
* Major abnormality of hepatic or renal function [ALT or AST >2-fold of the normal upper limit, creatinine > 1.5-fold- greater than the normal upper limit (excluding ALT > 1.5-fold greater than normal upper limit in patients with chronic stable hepatitis)]; concomitant infection with HBV and HCV;
* Hearing loss or clinically significant tinittus
* Use of inhaled or systemic antibiotics within 4 weeks prior to enrollment
* Needing oral or intravenous corticosteroids, or needing systemic corticosteroids within 30 days prior to enrollment
* Needing oral or intravenous anti-cholinergic medications, or needing systemic anti-cholinergic medications within 30 days prior to enrollment
* Needing long-term non-invasive mechanical ventilation or oxygen therapy (> 10 hrs daily) due to chronic respiratory failure
* Pregnancy or lactation
* Failure to understand or cooperate with the trial procedures
* Participation in other clinical trials within 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in sputum load of Pseudomonas aeruginosa at day 29 compared with baseline | 29 days
  Changes in sputum load of Pseudomonas aeruginosa at day 29 compared with baseline
Changes in Quality of Life in Bronchiectasis-Respiratory Symptom Score at day 29 compared with baseline | 29 days
  Changes in QoL-B-RSS at day 29 compared with baseline. The respiratory symptom domain contains 9 items describing patient's self assessment of her/his respiratory symptoms that affect the daily life. The total score for this domain is 100, with higher scores indicating better quality of life. No summation was made for the total score.

SECONDARY OUTCOMES:
The time to the first bronchiectasis exacerbation since randomization | 4 months
  The time to the first bronchiectasis exacerbation since randomization
The frequency of bronchiectasis exacerbation since randomization | 4 months
  The frequency of bronchiectasis exacerbation since randomization
The rate of isolation of Pseudomonas aeruginosa at day 85 | 85 days
  The rate of isolation of Pseudomonas aeruginosa at day 85
Changes in the load of Pseudomonas aeruginosa at day 85 compared with baseline | 85 days
  Changes in the load of Pseudomonas aeruginosa at day 85 compared with baseline
Changes in FEV1 pred% at days 29, 57 and 85 compared with baseline | 85 days
  Changes in the predicted % of forced expiratory volume in one second at days 29, 57 and 85 compared with baseline
Changes in 24-hour sputum volume at days 29, 57 and 85 compared with baseline | 85 days
  Changes in 24-hour sputum volume at days 29, 57 and 85 compared with baseline
Changes in sputum purulence at days 29, 57 and 85 compared with baseline | 85 days
  Changes in sputum purulence at days 29, 57 and 85 compared with baseline
Changes in Quality of Life in Bronchiectasis-Respiratory Symptom Score at day 85 compared with baseline | 85 days
  Changes in QoL-B-RSS at day 85 compared with baseline. The respiratory symptom domain contains 9 items describing patient's self assessment of her/his respiratory symptoms that affect the daily life. The total score for this domain is 100, with higher scores indicating better quality of life. No summation was made for the total score.
Changes in Bronchiectasis Health Questionnaire Sore at day 29 and 85 compared with baseline | 85 days
  Changes in BHQ Sore at day 29 and 85 compared with baseline. Theb BHQ contains 10 items, with higher scores indicating better quality of life. The total score was calculated as the weighted summation of the scores for the 10 individual items.
Peak and trough concentration of tobramycin at day 1 and 28 post-treatment | 29 days
  Peak and trough concentration of tobramycin at day 1 and 28 post-treatment
Changes in overall visual analogue scale at days 29 and 85 compared with baseline | 85 days
  Changes in overall VAS at days 29 and 85 compared with baseline. The VAS ranged from 0 to 10, with higher scores indicating poorer status. No summation of the score was made.
Changes in the minimal inhibitory concentration of Pseudomonas aeruginosa at days 29 and 85 compared with baseline | 85 days
  Changes in the MIC of Pseudomonas aeruginosa at days 29 and 85 compared with baseline (assessed with dilution methods for the sputum culture samples)

CONTACTS AND LOCATIONS:
Overall Officials: Nan-shan Zhong, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Wei-jie Guan, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Pasteur MC, Helliwell SM, Houghton SJ, Webb SC, Foweraker JE, Coulden RA, Flower CD, Bilton D, Keogan MT. An investigation into causative factors in patients with bronchiectasis. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1277-84. doi: 10.1164/ajrccm.162.4.9906120. PMID 11029331
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Aetiology of bronchiectasis in Guangzhou, southern China. Respirology. 2015 Jul;20(5):739-48. doi: 10.1111/resp.12528. Epub 2015 Mar 26. PMID 25819403
- [Background] Angrill J, Agusti C, De Celis R, Filella X, Rano A, Elena M, De La Bellacasa JP, Xaubet A, Torres A. Bronchial inflammation and colonization in patients with clinically stable bronchiectasis. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1628-32. doi: 10.1164/ajrccm.164.9.2105083. PMID 11719301
- [Background] Chalmers JD, Smith MP, McHugh BJ, Doherty C, Govan JR, Hill AT. Short- and long-term antibiotic treatment reduces airway and systemic inflammation in non-cystic fibrosis bronchiectasis. Am J Respir Crit Care Med. 2012 Oct 1;186(7):657-65. doi: 10.1164/rccm.201203-0487OC. Epub 2012 Jun 28. PMID 22744718
- [Background] Davies G, Wells AU, Doffman S, Watanabe S, Wilson R. The effect of Pseudomonas aeruginosa on pulmonary function in patients with bronchiectasis. Eur Respir J. 2006 Nov;28(5):974-9. doi: 10.1183/09031936.06.00074605. Epub 2006 Aug 9. PMID 16899482
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Li ZM, Zheng JP, Chen RC, Zhong NS. Effect of airway Pseudomonas aeruginosa isolation and infection on steady-state bronchiectasis in Guangzhou, China. J Thorac Dis. 2015 Apr;7(4):625-36. doi: 10.3978/j.issn.2072-1439.2015.04.04. PMID 25973228
- [Background] Wilson R, Aksamit T, Aliberti S, De Soyza A, Elborn JS, Goeminne P, Hill AT, Menendez R, Polverino E. Challenges in managing Pseudomonas aeruginosa in non-cystic fibrosis bronchiectasis. Respir Med. 2016 Aug;117:179-89. doi: 10.1016/j.rmed.2016.06.007. Epub 2016 Jun 7. PMID 27492530
- [Background] Orriols R, Hernando R, Ferrer A, Terradas S, Montoro B. Eradication Therapy against Pseudomonas aeruginosa in Non-Cystic Fibrosis Bronchiectasis. Respiration. 2015;90(4):299-305. doi: 10.1159/000438490. Epub 2015 Sep 5. PMID 26340658
- [Background] Hoppentocht M, Akkerman OW, Hagedoorn P, Alffenaar JW, van der Werf TS, Kerstjens HA, Frijlink HW, de Boer AH. Tolerability and Pharmacokinetic Evaluation of Inhaled Dry Powder Tobramycin Free Base in Non-Cystic Fibrosis Bronchiectasis Patients. PLoS One. 2016 Mar 9;11(3):e0149768. doi: 10.1371/journal.pone.0149768. eCollection 2016. PMID 26959239
- [Background] Bilton D, Henig N, Morrissey B, Gotfried M. Addition of inhaled tobramycin to ciprofloxacin for acute exacerbations of Pseudomonas aeruginosa infection in adult bronchiectasis. Chest. 2006 Nov;130(5):1503-10. doi: 10.1378/chest.130.5.1503. PMID 17099030
- [Background] Scheinberg P, Shore E. A pilot study of the safety and efficacy of tobramycin solution for inhalation in patients with severe bronchiectasis. Chest. 2005 Apr;127(4):1420-6. doi: 10.1378/chest.127.4.1420. PMID 15821224
- [Background] Drobnic ME, Sune P, Montoro JB, Ferrer A, Orriols R. Inhaled tobramycin in non-cystic fibrosis patients with bronchiectasis and chronic bronchial infection with Pseudomonas aeruginosa. Ann Pharmacother. 2005 Jan;39(1):39-44. doi: 10.1345/aph.1E099. Epub 2004 Nov 23. PMID 15562142
- [Background] Couch LA. Treatment With tobramycin solution for inhalation in bronchiectasis patients with Pseudomonas aeruginosa. Chest. 2001 Sep;120(3 Suppl):114S-117S. doi: 10.1378/chest.120.3_suppl.114s. PMID 11555565
- [Background] Orriols R, Roig J, Ferrer J, Sampol G, Rosell A, Ferrer A, Vallano A. Inhaled antibiotic therapy in non-cystic fibrosis patients with bronchiectasis and chronic bronchial infection by Pseudomonas aeruginosa. Respir Med. 1999 Jul;93(7):476-80. doi: 10.1016/s0954-6111(99)90090-2. PMID 10464834
- [Background] Barker AF, Couch L, Fiel SB, Gotfried MH, Ilowite J, Meyer KC, O'Donnell A, Sahn SA, Smith LJ, Stewart JO, Abuan T, Tully H, Van Dalfsen J, Wells CD, Quan J. Tobramycin solution for inhalation reduces sputum Pseudomonas aeruginosa density in bronchiectasis. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):481-5. doi: 10.1164/ajrccm.162.2.9910086. PMID 10934074
- [Derived] Guan WJ, Xu JF, Luo H, Xu XX, Song YL, Ma WL, Liang ZA, Liu XD, Zhang GJ, Zhang XJ, Li RK, Zhu SY, Zhang YJ, Cai XJ, Wei LP, Tian DB, Zhao H, Chen PY, Qu JM, Zhong NS; TORNASOL Study Group. A Double-Blind Randomized Placebo-Controlled Phase 3 Trial of Tobramycin Inhalation Solution in Adults With Bronchiectasis With Pseudomonas aeruginosa Infection. Chest. 2023 Jan;163(1):64-76. doi: 10.1016/j.chest.2022.07.007. Epub 2022 Jul 19. PMID 35863486